CLINICAL TRIAL: NCT03252470
Title: A Prospective, Post Market, Feasibility Study to Assess the Practical Utility of the OR BlackBox Platform When Used to Compare Surgical Technique During 2D Versus 3D Laparoscopic Bariatric Surgery
Brief Title: The BlackBox Study
Status: Completed | Type: Observational
Sponsor: Olympus Corporation of the Americas (Industry)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-SE-01
Record Dates: First submitted 2017-08-11; First posted 2017-08-17 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Laparoscopic Roux-en-y Gastric Bypass
Keywords: 2D laparoscopic surgery; 3D laparascopic surgery; laparoscopic roux-en-y gastric bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2D laparoscopic surgeries: Two-Dimensional Laparascopic Surgical Video System
  Interventions: Procedure: Laparoscopic Roux-en-y Gastric Bypass Surgery
- 3D laparoscopic surgeries: Three-Dimensional Laparascopic Surgical Video System
  Interventions: Procedure: Laparoscopic Roux-en-y Gastric Bypass Surgery

INTERVENTIONS:
Procedure: Laparoscopic Roux-en-y Gastric Bypass Surgery — Laparoscopic Roux-en-y Gastric Bypass Surgery

SUMMARY:
This is a hypothesis generating pilot study to compare the impact of 2D versus 3D visualization on surgical performance, as measured by the OR BlackBox platform, during laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Data published in 2008 estimated the global number of surgical procedures performed annually as 234 million with a rate of major perioperative complications reported between 3% and 17% in industrialized countries. As a derivative of these figures, it is estimated that approximately 7 to 40 million major complications occur worldwide each year. Studies have shown that between 39.6% and 54.2% of surgical complications occur in the operating room (OR); furthermore, it has been suggested that one third to half of all surgical errors are potentially avoidable. These findings have brought considerable attention to quality improvement in the technically demanding field of laparoscopic surgery wherein the risk of intraoperative error is increased by the sociotechnical complexity of the operative environment. In particular, there has been growing interest in evaluating surgical processes from a human factors point of view, as human factors, such as fatigue and mental workload, have become increasingly recognized as root causes of adverse surgical events and outcomes.

Among the most commonly reported errors in conventional laparoscopic surgery are technical errors associated with impaired depth perception; laparoscopic surgeons rely on two-dimensional (2D) video displays to guide their work in a three-dimensional (3D) space, resulting in the loss of depth perception and spatial orientation, as well as the experience of increased visual and cognitive load. Technical errors can be defined as manual errors of the surgeon (e.g. damage to adjacent structures) and procedural errors due to a lack of surgeon proficiency or experience. These errors are frequently described, especially when evaluating closed malpractice cases. These factors have been extensively examined but still remain controversial. A major limitation of error analyses of closed malpractice cases and root cause analyses of complications is the hindsight bias introduced through the knowledge of patient outcome.

Laparoscopic cameras with 3D display functionality were first developed in the early 1990s. The poor image quality produced by early cameras resulted in pronounced physical side effects, including dizziness, headache, and nausea; however, a significant technological advancement in the field of 3D laparoscopy has dramatically improved the usability of these systems. Despite these improvements and the potential for improved surgical safety, the use of 3D laparoscopic equipment remains limited in modern surgical centers. Outdated and conflicting research findings regarding the effectiveness of these systems and the physical side effects associated with their use may be contributing to slow adoption into clinical practice. Furthermore, investigations assessing the impact of 3D laparoscopy on surgical performance in the clinical setting are notably lacking. Thus, robust comparative evaluations of modern 2D and 3D laparoscopic surgical display systems in clinical settings are required to clearly elucidate the impact of 3D laparoscopy on surgical performance and safety with an aim to establish best practices in laparoscopic surgery.

The restoration of stereoscopic vision in laparoscopic surgery has the potential to mitigate these challenges and, to this end, the introduction of 3D stereoscopic displays in laparoscopic surgery may be beneficial to improving surgical safety. The purpose of this study is to compare the impact of 2D versus 3D visualization on surgical performance, as measured by the OR BlackBox Platform, during laparoscopic Roux-en-Y gastric bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Scheduled to undergo elective, primary roux-en-y gastric bypass surgery
3. BMI of 35 to 54.9
4. Willing and able to provide informed consent

Exclusion Criteria:

1. Previous open abdominal surgery
2. Previous open or laparoscopic upper GI surgery
3. Contraindicated for laparoscopic bariatric surgery
4. Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet all of the inclusion criteria and none of the exclusion criteria will be considered for enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Quantify operative performance and intraoperative errors | 12 months
  This pilot study will quantify operative performance and intraoperative errors after the introduction of the 2D and 3D technology using the following tools:
  * Generic Error Rating Tool (GERT)
  * Objective Structured Assessment of Technical Skill (OSATS)

SECONDARY OUTCOMES:
Significant adverse events | one month
  1. Clinically significant adverse events related to the device(s) and/or procedure

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Division of Surgery, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Informed Consent Form (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03252470/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03252470/Prot_SAP_001.pdf